CLINICAL TRIAL: NCT00512278
Title: Infliximab (Remicade®) as an Adjunct to Pegylated- Interferon α-2b and Ribavirin in the Treatment of Hepatitis C Virus Infection
Brief Title: Infliximab Treatment Along With Pegylated Interferon and Ribavirin in the Treatment of Hepatitis C
Acronym: PARTNER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nizar Zein (Other)
Collaborators: Centocor, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nizar Zein, Associate Professor of Medicine; Chief, Section of Hepatobiliary Diseases; Medical Director of Liver Transplantation, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PARTNER
Record Dates: First submitted 2007-08-03; First posted 2007-08-07 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Hepatitis C
Keywords: Hepatitis; HCV; Hepatitis C
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab (Experimental): Infliximab: 48 weeks of therapy with the combination of PEG INF-2b/RBV plus adjuvant infliximab
  Interventions: Drug: Infliximab
- Placebo (Placebo Comparator): Placebo: 48 weeks of therapy with Placebo and PEG INF-2b/RBV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Infliximab — Infliximab weight based injection at baseline, weeks 2,6,14,22,30,38,46
  Other Names: Remicade
  Arms: Infliximab
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The aim of the study is to investigate in subjects receiving their first course of peg-interferon α-2b plus ribavirin therapy for chronic HCV infection

DETAILED DESCRIPTION:
The aim of the study is to investigate in subjects receiving their first course of peg-interferon α-2b plus ribavirin therapy for chronic HCV infection (genotype 1) whether the addition of infliximab to a standard regimen of pegylated interferon α-2b in combination with ribavirin:

* increases the proportion of subjects attaining a sustained virological response SVR (undetectable blood Hepatitis C viral load 6 months after treatment)
* improves the safety profile compared to the same regimen without infliximab

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, >18 years of age with proven chronic (greater than 6 months) hepatitis C infection (genotype 1) who have never been treated with pegylated interferon α-2b and /or ribavirin.

Criteria for inclusion in this trial are as follows:

* Male or female, 18 years of age or older
* Positive HCV RNA, Genotype 1, treatment naïve (never received pegylated interferon and / or ribavirin)
* Evidence of chronic HCV infection for at least six months prior to screening
* Findings on liver biopsy within the past 36 months that are consistent with the presence of chronic hepatitis C infection.
* Negative hepatitis B surface antigen
* No evidence of hemochromatosis
* Hemoglobin ≥12 g/dL for females and ≥13 g/dL for males
* WBC ≥3.0 x 109/L and neutrophils ≥1.5 x 109/L
* Platelets ≥80 x109/L
* Direct Bilirubin WNL +/- 50% of central laboratory normal range. Total bilirubin ≤1.6.
* Albumin within normal limits
* Serum creatinine within normal limits.
* Serum thyroid stimulating hormone (TSH) levels within normal limits
* Men and women of childbearing potential must use two forms of adequate birth control measures for the duration of the study and should continue such precautions for 6 months after receiving the last infusion.
* Subjects with a history of mild depression may be considered for entry into this study.
* No history of latent or active TB.

Exclusion Criteria:

* Women who are pregnant, nursing, or planning pregnancy within 6 months after the last infusion and men with partners who are pregnant at baseline or intend to become pregnant within 6 months after the last infusion.
* Known allergy against infliximab, ribavirin, or pegylated interferon
* Decompensated liver disease characterized as decreased hepatic synthetic functioning with abnormal albumin and bilirubin levels, prolonged prothrombin time or complications including ascites or recent variceal bleeding
* have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidiomycosis (Valley Fever)
* History of autoimmune hepatitis or a history of poorly controlled autoimmune disease
* Use of other systemic anti-inflammatory medication except NSAIDs and low dose systemic steroids
* Previous treatment with monoclonal antibodies or antibody fragments
* History of receiving human/murine recombinant products or a known allergy to murine products
* Documentation of seropositive for human immunodeficiency virus (HIV)
* History of alcohol or substance abuse within the preceding 6 months that, in the opinion of the investigator, may increase the risks associated with study participation or study agent administration, or may interfere with interpretation of results
* History of serious infections (e.g., hepatitis, pneumonia or pyelonephritis) in the previous 3 months
* Opportunistic infection within 6 months prior to screening
* History of lymphoproliferative disease
* Currently have any known malignancy or have a history of malignancy within the previous 5 years, with the exception of basal cell or squamous cell carcinoma of the skin that has been fully excised with no evidence of recurrence
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, or cerebral disease
* Treatment with any other therapeutic agent targeted at reducing TNF within 3 months of screening
* Presence of a transplanted solid organ
* Concomitant diagnosis or history of congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nizar N Zein, MD, Principal Investigator — The Cleveland Clinic
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Center for Liver Disease and Transplantation, Los Angeles, California
  - Advanced Medical Research Center, Port Orange, Florida
  - University of Louisville, Louisville, Kentucky
  - Case Medical Center, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Brooke Army Medical Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment 2007-2011 Data Lock Nov 22, 2012 Sites
  1. The Cleveland Clinic
  2. University Hospitals of Cleveland
  3. Cedar Sinai Medical Center, Los Angeles,
  4. The Liver Institute at Methodist Dallas
  5. Brooke Army Medical Center, San Antonio
  6. Advanced Medical Research Center, Daytona Beach.
  7. University of Louisville, Louisville
Pre-assignment Details: 220 subjects screened and 149 randomized Reasons for exclusion were multiple including malignancy, liver failure, negative HCV RNA, abnormal lab values, poorly controlled diabetes, psych disorders, positive tuberculosis skin test, seizure disorder, inability to get labs or liver biopsy, pregnancy, patient declining, other (cardiomypathy, MS, etc.)
Groups:
- A Infliximab: Infliximab: 48 weeks of therapy with the combination of PEG INF-2b/RBV plus adjuvant infliximab
  Infliximab : Infliximab weight based injection at baseline, weeks 2,6,14,22,30,38,46
  All patients received triple therapy (pegylated interferon (PEG IFN)/ribavirin/infliximab) at approved doses
- B Placebo: Placebo: 48 weeks of therapy with Placebo and PEG INF-2b/RBV
  Placebo : Placebo
  All patients received triple therapy (pegylated interferon (PEG IFN)/ribavirin/placebo) at approved doses. Placebo infusions were timed similar to infliximab for patients in arm A of the study
Period: Overall Study
Arm/Group | A Infliximab | B Placebo
Started | 73 | 73
Completed | 45 | 56
Not Completed | 28 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A Infliximab | B Placebo | Total
Number analyzed (Participants) | 73 | 73 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 73 | 73 | 146
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (9.78) | 47.2 (9.38) | 46.9 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 40 | 42 | 82
Region of Enrollment [Number; unit: participants]
  United States | 73 | 73 | 146

OUTCOME MEASURES:

1. Primary Outcome: A Comparison of the Percentage of Chronic Hepatitis C Subjects (Treatment Naive,Genotype 1) Who Achieve SVR at Week 72, After 48 Weeks of Treatment.
Description: A comparison of the Proportion of Chronic Hepatitis C Subjects (Treatment Naive,Genotype 1) Who Achieve SVR at Week 72, After 48 Weeks of TreatmentSVR in both study arms
Time Frame: 72 Weeks from initiation of treatment
Population: Included all patients who received at least one dose of treatment in both study arms
Measure: Number; unit: percentage of participants
Arm/Group | A Infliximab | B Placebo
Number analyzed (Participants) | 73 | 73
percentage of participants | 28.8 | 31.5
Statistical Analysis 1: Comparison: A Infliximab vs B Placebo; Test type: Non-Inferiority or Equivalence — Assuming a 25% difference in the rate of SVR between the PEG INF/RBV plus infliximab group (70%) and the PEG INF/RBV (45%) group, a power of 0.85 and an alpha level of 0.05, 75 patients for each group was estimated; p = 0.718, t-test, 2 sided

2. Secondary Outcome: A Comparison of the Percentage of Participants With Non-detectable HCV-RNA After 24 Weeks of Therapy.
Description: A comparison of the proportion of the subject population with non-detectable HCV-RNA after 24 wks of therapy.
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Groups:
- A Infliximab: Infliximab: 48 weeks of therapy with the combination of PEG INF-2b/RBV plus adjuvant infliximab
  Infliximab : Infliximab weight based injection at baseline, weeks 2,6,14,22,30,38,46
  All patients recieved triple therapy (pegylated interferon (PEG IFN)/ribavirin/infliximab) at approved doses
- B Placebo: Placebo: 48 weeks of therapy with Placebo and PEG INF-2b/RBV
  Placebo : Placebo
  All patients recieved triple therapy (pegylated interferon (PEG IFN)/ribavirin/placebo) at approved doses. Placebo infusions were timed simialr to infliximab for patients in arm A of the study
Arm/Group | A Infliximab | B Placebo
Number analyzed (Participants) | 73 | 73
Participants | 40 | 41

3. Primary Outcome: Number of Participants Achieving Sustained Virological Response (SVR)
Description: HCV RNA negativity at 24 weeks after completion of all study medications
Time Frame: 24 weeks after completion of all study medications
Measure: Count of Participants; unit: Participants
Arm/Group | A Infliximab | B Placebo
Number analyzed (Participants) | 73 | 73
Participants | 21 | 23
Statistical Analysis 1: Comparison: A Infliximab vs B Placebo; SVR was the primary outcome to calculate sample size. Assuming a 25% difference in the rate of SVR between the the two groups, a power of 0.85 and an alpha level of 0.05, 75 patients for each group was estimated. This analysis included patients randomized and received at least one dose of study drugs. A 2-sided probability value of < 0.05 was considered statistically significant. Univariate and multivariable logistic regression were used for factors associated with an SVR; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.718, t-test, 2 sided — Univariate and multivariable logistic regression were used for factors associated with an SVR

4. Secondary Outcome: Percentage of Participants Experiencing Serious Adverse Events
Description: The severity of adverse events was graded according to modified World Health Organization grades as mild, moderate, severe, or life-threatening
Time Frame: 72 Weeks from initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | A Infliximab | B Placebo
Number analyzed (Participants) | 73 | 73
Participants | 21 | 13

5. Secondary Outcome: Percentage of Participants Experiencing Medically Significant Infections
Description: Medically significant infection was defined as an infection requiring the use of intravenous antibiotics or hospitalization.
Time Frame: 72 weeks from initiation of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | A Infliximab | B Placebo
Number analyzed (Participants) | 73 | 73
Participants | 10 | 3

ADVERSE EVENTS:
Time Frame: 72 weeks
Arm/Group | A Infliximab | B Placebo
All-Cause Mortality (participants affected / at risk) | 0/73 | 1/73
Serious Adverse Events (participants affected / at risk) | 21/73 | 13/73
Other Adverse Events (participants affected / at risk) | 73/73 | 73/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A Infliximab (N=73) | B Placebo (N=73)
Anemia (Blood and lymphatic system disorders) | 4 | 2 — hemoglobin less than 8.5g/dL
Medically Significant Infections (Infections and infestations) | 10 | 3
Coordination Abnormal (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 3
Severe Dehydration (General disorders) | 3 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0
Chest Pain (General disorders) | 1 | 0 — Etiology not determined.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A Infliximab (N=73) | B Placebo (N=73)
Fatigue (General disorders) | 55 | 54
Influenza-Like Illness (General disorders) | 23 | 17
Irritability (General disorders) | 20 | 21
Pyrexia (General disorders) | 21 | 26
Chills (General disorders) | 13 | 28
Nausea (Gastrointestinal disorders) | 36 | 41
Diarrhea (Gastrointestinal disorders) | 11 | 23
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 26
Rash (Skin and subcutaneous tissue disorders) | 29 | 23
Alopecia (Skin and subcutaneous tissue disorders) | 18 | 17
Any Infection (Infections and infestations) | 48 | 42
Headache (Nervous system disorders) | 42 | 39
Dizziness (Nervous system disorders) | 14 | 16
Insomnia (Psychiatric disorders) | 31 | 27
Depression (Psychiatric disorders) | 21 | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 39 | 25
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 27
Anemia (Blood and lymphatic system disorders) | 19 | 19
Neutropenia (Blood and lymphatic system disorders) | 10 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No